CLINICAL TRIAL: NCT00338455
Title: Investigation of the Use of Natrecor (Nesiritide) in Transplant-Eligible Management of Congestive Heart Failure-TMAC
Brief Title: Natrecor (Nesiritide) in Transplant-Eligible Management of Congestive Heart Failure-TMAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMC acknowledged no safety concerns with the trial, recommending that the trial be terminated due to slow enrollment
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR003649; A051; TMAC
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Congestive Heart Failure; Cardiac Transplantation; Renal Insufficiency; Renal Failure
Keywords: Congestive heart failure; cardiac transplantation; renal insufficiency; renal failure; dialysis; ultrafiltration; vasodilator; Natrecor (nesiritide)
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain; Milrinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): Natrecor (nesiritide)+Standard Care+dobutamine or milrinone 28-day continuous infusion no bolus 3-hour 0.005 mcg/kg/min may be titrated to 0.015 mcg/kg/min
  Interventions: Drug: Natrecor (nesiritide)+Standard Care+dobutamine or milrinone
- 002 (Placebo Comparator): Placebo+Standard Care+dobutamine or milrinone 28-day continuous infusion no bolus 3-hour 0.005 mcg/kg/min may be titrated to 0.015 mcg/kg/min
  Interventions: Drug: Placebo+Standard Care+dobutamine or milrinone

INTERVENTIONS:
Drug: Natrecor (nesiritide)+Standard Care+dobutamine or milrinone — 3-hour 0.005 mcg/kg/min, may be titrated to 0.015 mcg/kg/min
  Arms: 001
Drug: Placebo+Standard Care+dobutamine or milrinone — 28-day continuous infusion, no bolus
  Arms: 002

SUMMARY:
The purposes of this study in United Network for Organ Sharing (UNOS) Status 1B (or country equivalent) cardiac transplant candidates are to assess the safety and efficacy of Natrecor (nesiritide). The study will evaluate the drug's ability to prevent clinical worsening when administered as a 28-day continuous intravenous infusion in patients receiving standard care and continuous intravenous infusion of dobutamine or milrinone.

DETAILED DESCRIPTION:
Endogenous B-type natruretic peptide (BNP) concentrations correlate with heart failure (HF) severity and are significantly elevated in severe end-stage HF patients. However, normal biologic compensatory responsiveness to BNP is attenuated in patients with severe HF. Patients who are UNOS 1B cardiac transplant candidates have relatively few options for therapy, despite the fact that they constitute a very ill patient population. These options include getting a transplant, if one is available, receiving intravenous inotropes and/or vasodilators, or being implanted with a circulatory support device (e.g. Left Ventricular Assist Device). Natrecor (Nesiritide) is a human recombinant form of BNP approved for use in the treatment of acute decompensated HF. Limited information is available from controlled clinical trials on the effects of Natreor (nesiritide) infusion for longer than 72 hours. However, based on reports in the literature, Natrecor (nesiritide) has been used by independent investigators for much longer durations in end-stage HF patients, including UNOS Status 1B cardiac transplant candidates, who are refractory to standard care. In these patients, Natrecor (nesiritide) has been safely administered by continuous infusion for more than 2 and up to 210 days. These experiences showed that continuous Natrecor (nesiritide) infusion was well tolerated, uniformly improved hemodynamics (circulation of the blood and the forces involved), maintained stable renal (kidney) function, and reduced the need for ventricular assist devices during the prolonged wait for heart transplant. In controlled clinical trials reported in literature, Natrecor (nesiritide) was given concomitantly with several other standard HF therapeutic agents, such as diuretics, angiotensin-converting enzyme (ACE) inhibitors, beta-blockers, dopamine, dobutamine, anticoagulants, digoxin, and oral nitrates. Concomitant dosing was well tolerated, and no drug interactions were observed. No randomized controlled trial has been conducted to evaluate the safety of combination nesiritide and milrinone therapy. Several investigations were undertaken because of concerns over the potential additive hypotensive (lowering blood pressure) effect that these two agents may exert when administered concurrently. The study investigators reported that concurrent dosing of milrinone and nesiritide appeared to be safe and beneficial, without evidence of an additive hypotensive (lowering blood pressure) effect. The TMAC trial will investigate the safety and efficacy of Natrecor (nesiritide), compared with placebo, when added to standard care in the management of end-stage refractory HF.This prospective, randomized(patients are assigned different treatments based on chance), parallel, multicenter, double-blind (neither the doctor nor the patient knows whether the patient is being administered a placebo or the test drug), placebo-controlled study will be conducted with UNOS Status 1B (or equivalent) cardiac transplant candidates who are receiving standard care and continuous IV infusion of dobutamine or milrinone while awaiting heart transplantation. Approximately 120 patients will participate in this study. Enrolled patients will be randomized 1:1 to receive Natrecor (nesiritide) by continuous infusion in addition to standard care and one inotrope (drugs such as dobutamine or milrinone used to increase the heart rate and improve the force of cardiac contraction), or to receive placebo by continuous infusion in addition to standard care and one inotrope (dobutamine or milrinone). Patients will be managed as inpatients or outpatients, according to the guidelines in this protocol and study center practices. All patients will continue to receive their usual long-term cardiac medications (excluding commercial nesiritide). Study drug dose adjustments may be made according to the guidelines in this protocol and the investigator's clinical judgment, and in accordance with the dosing guidelines.Study drug will be administered as a continuous intravenous infusion under the control of a programmable ambulatory infusion pump for the 28-day treatment period. Patients will be hospitalized for study drug initiation and titration to ensure safety, observe tolerability, and achieve the recommended study drug dose. Day 0 (Screening) will entail completing required procedures and randomization. Baseline and screening procedures may occur on the same day. A window of up to 7 days will be permitted between Day 0 (Screening) and Day 1 (Baseline) visits if circumstances delay initiation of study drug dosing. The following day, Day 1 (Baseline), continuous infusion of study drug will begin. Patients will be hospitalized for a minimum of 3 days after starting the study drug for titration and dose optimization. A dose optimization period of up to 5 days will be permitted. Patients will be eligible for discharge following completion of the study procedures on the 4th dosing day (Day 4). Patients will return to the clinic for weekly visits (± 2 days) through Day 28 (Termination of Treatment) and again at Day 35 for a 7-day post dosing safety visit. On the Day 28 visit (Termination of Treatment), Patients may be hospitalized for up to 24 hours at the investigator's discretion to undergo end of treatment study procedures. This study includes two substudies: the Pulmonary Function Testing Substudy and the Glomerular Filtration Rate Substudy. All TMAC Patients will be asked to participate in these substudies. Participation is optional and does not affect enrollment or participation in TMAC. The Study Hypothesis is that continuous administration of Natrecor (nesiritide) over 28 days when added to standard care (including inotropes) is safe and provides a clinical benefit when compared to placebo added to standard care (including inotropes) therapy. Study drug will be administered continuously as a fixed-rate infusion for 28 days without a bolus dose. Natrecor (nesiritide) dosing will begin at 0.005 mcg/kg/min and may be titrated to a maximum dose of 0.015 mcg/kg/min.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for a United Network for Organ Sharing (UNOS) Status 1B heart transplant candidate, or, if outside the US, have comparable status
* must also be a primary transplant candidate waiting to receive a single cardiac allograft
* must be receiving continuous intravenous infusion of dobutamine or milrinone through a double-lumen central catheter or a double-lumen percutaneously inserted central catheter for at least 3 consecutive days before randomization
* must be willing and able to participate in the study assessments and follow up procedures
* male and female subjects of childbearing potential agree to use two highly effective methods of birth control for the duration of the study.

Exclusion Criteria:

* Not have systolic blood pressure (SBP) consistently < 80 mm Hg, or have clinically significant orthostatic hypotension
* not weigh > 130 kg
* not have a ventricular assist device (VAD), or anticipate the need for a VAD, during the 28-day study drug treatment period
* not have received placement of an internal cardiac defibrillator (ICD) or external cardiac defibrillator (ECD) within 72 hours before randomization
* not require chronic hemodialysis or peritoneal dialysis to treat renal failure, or had acute dialysis or ultrafiltration within 7 days before randomization
* not have received antibiotic treatment within 7 days before randomization-antibiotics are permissible for any prophylactic use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.
Locations (14):
- United States (14):
  - Stanford, California
  - Tampa, Florida
  - Chicago, Illinois
  - Maywood, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - New York, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 16 participants randomized in the study, 1 participant randomized to receive nesiritide was not administered study drug due to investigator decision.Summaries of baseline characteristics are based on the 16 participants who were randomized in the study. Safety and efficacy analyses were based on the 15 participantswho received study drug.
Groups:
- Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone: Nesiritide - 28-day continuous infusion, no bolus; 3-hour 0.005 mcg/kg/min, may be titrated to 0.015 mcg/kg/min.
- Placebo + Standard Care + Dobutamine or Milrinone: Placebo - 28-day continuous infusion, no bolus; 3-hour 0.005 mcg/kg/min, may be titrated to 0.015 mcg/kg/min.
Period: Overall Study
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Started | 9 | 7
Administered Study Drug | 8 | 7
Completed | 6 | 6
Not Completed | 3 | 1
Not completed — Death | 2 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.80) | 54.6 (4.65) | 53.1 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 4 | 12
Glomerular Filtration Rate (GFR) [Number; unit: Participants] — Estimate of the GFR using serum creatinine and demographic factors.
  Participants
    GFR < 60 | 4 | 4 | 8
    GFR > = 60 | 5 | 3 | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (5.53) | 31.7 (5.79) | 30.5 (5.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive Without Renal, Hemodynamic, or Electrical Clinical Worsening Through Day 28 (Termination of Treatment)
Description: Number of calendar days alive without renal, hemodynamic, or electrical clinical worsening through Day 28 (termination of treatment or early discontinuation of treatment, whichever occurred first). The endpoint was not normalized for time on study.
Time Frame: 28 days
Population: Early termination of the study due to enrollment difficulties; efficacy not analyzed.
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Changes in Pulmonary Capillary Wedge Pressure (PCWP)
Time Frame: 28 days
Population: Early termination of the study due to enrollment difficulties; efficacy not analyzed.
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: All Cause Mortality
Time Frame: Day 30 and Months 2 and 6
Population: Early termination of the study due to enrollment difficulties; efficacy not analyzed.
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in Pulmonary Artery Pressure (PAP): Systolic, Diastolic, and Mean
Time Frame: 28 days
Population: Early termination of the study due to enrollment difficulties; efficacy not analyzed.
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety evaluations were to be performed on treatment and at Months 2 and 6.
Arm/Group | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone | Placebo + Standard Care + Dobutamine or Milrinone
Serious Adverse Events (participants affected / at risk) | 4/8 | 3/7
Other Adverse Events (participants affected / at risk) | 7/8 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone (N=8) | Placebo + Standard Care + Dobutamine or Milrinone (N=7)
sepsis (Infections and infestations) | 1 | 0
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pneumonia (Infections and infestations) | 1 | 0
cardiac failure congestive (Respiratory, thoracic and mediastinal disorders) | 3 | 1
cardiac failure (Cardiac disorders) | 0 | 1
gastroenteritis (Infections and infestations) | 1 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
anaphylactic reaction (Immune system disorders) | 0 | 1
convulsion (Nervous system disorders) | 0 | 1
staphylococcal sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natrecor (Nesiritide)+Standard Care+Dobutamine or Milrinone (N=8) | Placebo + Standard Care + Dobutamine or Milrinone (N=7)
gout (Metabolism and nutrition disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 2 | 1
constipation (Gastrointestinal disorders) | 1 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
oedema peripheral (General disorders) | 1 | 1
hypotension (Vascular disorders) | 1 | 1
catheter site infection (Infections and infestations) | 1 | 0
clostridial infection (Infections and infestations) | 1 | 0
clostridium colitis (Infections and infestations) | 1 | 0
naospharyngitis (Infections and infestations) | 0 | 1
staphylococcal infection (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 1
catheter related complication (General disorders) | 1 | 0
catheter site discharge (General disorders) | 1 | 0
rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
erythema (Skin and subcutaneous tissue disorders) | 0 | 1
deep vein thrombosis (Vascular disorders) | 1 | 0
jugular vein distension (Vascular disorders) | 0 | 1
blood creatinine increased (Investigations) | 1 | 0
blood glucose increased (Investigations) | 0 | 1
gallop rythm present (Investigations) | 1 | 0
hepatomegaly (Hepatobiliary disorders) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 1 | 0
hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
dyspepsia (Gastrointestinal disorders) | 0 | 1
post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
depression (Psychiatric disorders) | 1 | 0
insomnia (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination of the study due to enrollment difficulties (change in standard of care for patient population as well as changing organ allocation rules by United Network for Organ Sharing); efficacy not analyzed due to limited sample size (n=16).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days